CLINICAL TRIAL: NCT00317616
Title: The Pre-symptomatic Familial Amyotrophic Lateral Sclerosis (Pre-fALS) Study
Acronym: Pre-fALS
Status: Recruiting | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: ALS Association (Other)
Responsible Party: Principal Investigator, Michael Benatar, Professor, University of Miami
Other Study IDs: Pre-fALS
Record Dates: First submitted 2006-04-24; First posted 2006-04-25 (Estimated); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: FALS; SOD1; familial; genetic testing; genetic counseling; ALS; C9ORF72; TARDBP; VCP; FUS; PFN1
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Frontotemporal Dementia With Motor Neuron Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma, CSF, DNA, Urine, Cell lines
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Unaffected individuals from families in which the genetic cause of ALS is known: This population would include pre-symptomatic individuals at genetic risk for ALS or a related neurodegenerative disorder (i.e., FTD).

SUMMARY:
Pre-fALS is a prospective natural history and biomarker study of people not yet affected with ALS, but who are at genetic risk for developing ALS. The investigators aim to recruit unaffected (healthy) people from familial ALS (fALS) pedigrees in which a known genetic mutation associated with ALS has been identified; for this study, a fALS pedigree is one with two biologically related individuals who have or have had ALS and/or FTD. Individuals who may be at genetic risk for ALS and who belong to families with at least one affected family member who has tested positive for a known ALS genetic mutation may also be eligible to participate. Our goal is to study the pre-symptomatic phase, onset and progression of ALS and to learn more about genetic and environmental factors that put people at risk for developing ALS.

DETAILED DESCRIPTION:
Healthy individuals from fALS families with a known genetic mutation will be included in this study. We encourage people who have previously undergone genetic testing and were found to carry the mutation that affects their family as well as those who do not know their genetic status to contact us. Those who wish to participate and to learn the results of genetic testing, may do so after undergoing genetic counseling. It is also possible to participate without learning the results of genetic testing. Participants eligible to complete study visits will travel to Miami (at our expense) approximately every 12-24 months for a period of 10 years or longer and will perform various biomarker procedures. Between visits, participants will complete phone calls about their health.

ELIGIBILITY:
Inclusion Criteria

* A member of a family in which a mutation in a gene associated with ALS has been identified.
* No symptoms to suggest the presence of ALS (i.e. study participants must currently be healthy).
* Having at least 50% probability of carrying an ALS associated gene mutation based on family pedigree.
* Willingness to undergo genetic testing, with the option of whether or not to learn the results.
* Willingness and availability to travel to Miami for a few days approximately every 12 to 24 months to complete biomarker procedures (e.g, MRI, blood draws, spinal tab/lumbar puncture, cognitive testing)

Exclusion Criteria

* Diagnosis of ALS
* Any condition or situation which, in the PI's opinion, could confound the biomarker data or may interfere with the individual's participation and compliance with the study protocol, including but not limited to neurological, psychological and/or medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy individuals who harbor a mutation in a gene associated with ALS.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2006-04; Primary Completion 2037-12 (Estimated); Study Completion 2037-12 (Estimated)

PRIMARY OUTCOMES:
Risk Factors for Progression to familial ALS | Years

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Benatar, MD, PhD., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No